CLINICAL TRIAL: NCT02156219
Title: Building Capacity of State and Local Actors to Respond to Violence Against Women: Impact Evaluation of Separating Women and Men in the Metro of Mexico City, Component of the Program "Viajemos Seguras"
Brief Title: Impact Evaluation of Separating Women and Men in the Metro of Mexico City
Status: Suspended | Type: Observational
Why Stopped: The STC has had financial limitations to start implementing the intervention.
Sponsor: Econometría Consultores (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Other Study IDs: ATN/MG-13064-RG ECO577-1
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-02

CONDITIONS: Violence Against Women (VAW)
MeSH Terms: interventions — Menogaril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Under separation: Exposure to the separation of women and men in the metro of Mexico City.
  Interventions: Other: Separation of women and men in the metro of Mexico City
- No treatment: Non exposure to the separation of women and men in the metro of Mexico City.

INTERVENTIONS:
Other: Separation of women and men in the metro of Mexico City — The measure of separation between men and women exists in all modes of public transport in Mexico City (metro, metro-bus, trolley, bus and light rail), although it is not 100% implemented on all lines and in all hours. These differences in implementation schedule can be a way to identify a treatment group and a control group, and the fact that it has not been implanted in all lines/paths will allow to have a baseline.
  The implementation of the measure of separation of men and women on the subway consists of three operational tasks:
  1. Control: Surveillance that men do not use cars corresponding to women.
  2. Dosage: Regulation of entry women.
  3. Assignment: Of the women, to the part of the platform where the first wagons stop.
  Groups: Under separation

SUMMARY:
The purpose of this study is to determine whether the separation of men and women in the metro of Mexico City leads to an improvement in the violence and perception of violence towards women.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the separation of men and women in the metro of Mexico City leads to an improvement in the violence and perception of violence towards women.

The separation of men and women will take place in the Line 5 of the metro system. The separation will operate between 6:00am-10:00am and 2:00pm and 10:30pm. Line 4 and 6 will be used to estimate the counterfactual.

Women eligible to participate in the study will be those aged 18 and 65 years who use lines 4, 5, and 6 between 7am and 9am or between 11am and 1pm before the separation between men and women is implemented. Eligible women must reside in Mexico City or the metropolitan area of the Valley of Mexico (60 municipalities agglomerates in the State of Hidalgo and Mexico State).

Women will be recruited in the metro before the separation between men and women is implemented. They will be asked for their name, e-mail and telephone number. Also before the separation is implemented, they will be asked to answer a telephone survey to collect baseline information. The same women will be contacted again in the following 12 to 15 months to collect the endline survey, also by phone. The implementation of the separation will take place after the baseline survey has been collected.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 who reside in Mexico City or the metropolitan area of the Valley of Mexico and that are users on the Metro lines 4, 5 and 6 between 7 and 9 or 11 and 1pm at baseline

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18-65 who reside in Mexico City or the metropolitan area of the Valley of Mexico and that are users on the Metro lines 4, 5 and 6 between 7 and 9 or 11 and 1pm at baseline
Sampling Method: Non-Probability Sample
Enrollment: 2360 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Perception of safety in public transport | Average of 1 year since the start of the intervention
  The outcome will be measure through a survey to women who use the lines 4, 5 and 6 of the metro system of Mexico City.

SECONDARY OUTCOMES:
Events of Violence against women in public transport | 6 months
  The outcome will be measure through a survey to women who use the lines 4, 5 and 6 of the metro system of Mexico City.
Behaviors, attitudes and perceptions of women about violence in public transport | Average of 1 year since the start of the intervention
  The outcome will be measure through a survey to women who use the lines 4, 5 and 6 of the metro system of Mexico City.
Women's autonomy (economic performance, activities outside the home) | Average of 1 years since the start of the intervention
  The outcome will be measure through a survey to women who use the lines 4, 5 and 6 of the metro system of Mexico City.
Negative externalities (perception of safety outside the public transport) | 6 months
  The outcome will be measure through a survey to women who use the lines 4, 5 and 6 of the metro system of Mexico City.

CONTACTS AND LOCATIONS:
Locations (1):
- Econometria Consultores, Bogotá, Colombia